CLINICAL TRIAL: NCT01613261
Title: A Multicenter, Open-label, Phase 1b Study of TAK-733 (an Oral MEK Inhibitor) in Combination With Alisertib (an Oral Aurora A Kinase Inhibitor) in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: Study of TAK-733 in Combination With Alisertib in Adult Patients With Advanced Nonhematologic Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20002; 2012-000831-22 (EudraCT Number)
Record Dates: First submitted 2012-06-01; First posted 2012-06-07 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Nonhematologic Malignancies
Keywords: TAK-733,; alisertib,; MLN8237,; Oral MEK Inhibitor,; Oral Aurora A Kinase Inhibitor
MeSH Terms: interventions — TAK 733; MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-733 and alisertib (Experimental)
  Interventions: Drug: TAK-733 and alisertib

INTERVENTIONS:
Drug: TAK-733 and alisertib — TAK-733 will be administered orally once daily (QD) on Days 1 through 14 of the 21-day cycle.
  Alisertib will be administered orally twice daily (BID) on Days 1 through 7 of the 21-day cycle.

SUMMARY:
This is a Multicenter, Open-label, Phase 1b Study of TAK-733 in Combination With Alisertib in Adult Patients With Advanced Nonhematologic Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Patients must have a diagnosis of a solid tumor malignancy for which standard, curative, or life-prolonging treatment does not exist or is no longer effective
* Radiographically or clinically evaluable tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Female patients who are post menopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 30 days after the last dose of study drug or agree to abstain from heterosexual intercourse
* Male patients who agree to practice effective barrier contraception through 4 months after the last dose of alisertib or agree to abstain from heterosexual intercourse
* Voluntary written consent
* Clinical laboratory values as specified in the protocol

Exclusion Criteria:

* Female patients who are breastfeeding and lactating or pregnant
* Serious medical or psychiatric illness or laboratory abnormality that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Treatment with any investigational products within 28 days before the first dose of study drug
* Prior treatment with Aurora A-targeted agents, including alisertib
* Prior treatment with MEK inhibitors, including TAK-733
* Prior treatment with BRAF inhibitors
* Systemic anticancer therapy within 21 days before the first dose
* Prior biologic or immunotherapy within 28 days before the first dose
* Major surgery or serious infection within 14 days before the first dose
* Life-threatening illness unrelated to cancer
* Known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C
* Cardiac condition as specified in study protocol or severe CNS, pulmonary, renal or hepatic disease
* Known GI conditions or GI procedure that could interfere with the oral absorption or tolerance of study drugs
* History of uncontrolled sleep apnea syndrome or other conditions that could result in excessive daytime sleepiness
* History of ongoing or a newly diagnosed eye abnormality
* Symptomatic brain metastases

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs), assessments of clinical laboratory values, and vital sign measurements | From signing of the informed consent form through 30 days after the last dose of study drug
  To evaluate the safety profile and to determine DLTs, MTDs, and RP2D of oral TAK-733 + alisertib in patients with advanced nonhematologic malignancies
TAK-733 and alisertib PK parameters including, but not limited to Cmax, Tmax, Area Under Curve (AUC), apparent oral clearance (CL/F), peak-to-trough ratio, and accumulation ratio | Escalation and MTD Refinement: Cycle 1-Day 1, 2, 7, 8, 14,and 15; Tumor Expansion Cohort: Cycle 1-Day 1, 7, 8, and 15; Cycle 2-Day 1, 8,and 15; PK Expansion Cohort: Cycle 1-Day 1, 7, and 8; Cycle 2-Day 7, 14, and 15. Each cycle is a 21 days cycle
  To characterize the single- and multiple-dose plasma PK of TAK-733 and alisertib in patients with advanced nonhematologic malignancies

SECONDARY OUTCOMES:
Measures of disease response, including objective response rate and duration of response based on investigator's assessment using RECIST guidelines | On screening; Cycle 2: between Day 15 and 21, and every third cycle thereafter (5,8,11 etc.) until progressive disease for approximately 1 year
  To evaluate evidence of antitumor activity of TAK-733 + alisertib

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- South Texas Accelerated Research Therapeutics (START), San Antonio, Texas, United States